CLINICAL TRIAL: NCT02356510
Title: Which One Should be Treated in the Setting of Acute ST Elevation Myocardial Infarction - Culprit Lesion or Culprit Vessel?
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ugur ARSLAN, Associate Proffessor of Cardiology, Head of Department, Samsun Education and Research Hospital
Other Study IDs: SamsunERH
Record Dates: First submitted 2015-02-01; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; TIMI flow; culprit lesion; culprit vessel
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Culprit lesion: Patients who underwent culprit lesion only PCI during primary intervention
  Interventions: Procedure: Primary PCI
- Culprit vessel: Patients who underwent culprit lesion only PCI during primary intervention
  Interventions: Procedure: Primary PCI

INTERVENTIONS:
Procedure: Primary PCI

SUMMARY:
The current guidelines still recommend emergent PCI of the culprit lesion and state that primary PCI should be limited to the culprit vessel with the exception of cardiogenic shock and persistent ischaemia after PCI of the supposed culprit lesion. This recommendation is based on a high number of studies. However, several studies are present about the safety and efficacy of non-culprit vessel PCI during acute MI. Nowadays, the debate is increasingly going on about the PCI of the non-culprit arteries during the index event with newer prospective randomized studies. Besides, it is still unclear for the culprit artery whether to treat only the culprit lesion or all the other lesions in the culprit vessel during the index event. The present report describes a retrospective comparison between the two strategies during primary PCI for STEMI, looking for their influence on the clinical and angiographic course of the patients.

DETAILED DESCRIPTION:
Patient selection: This multi-centre retrospective study included patients from 3 high-volume primary PCI centres in Turkey. A total number of 5512 patients underwent emergent PCI for acute STEMI between January 2011 and December 2013. From this patient population, patients were looked for the presence of an additional lesion to the culprit lesion (CL). Additional lesion was defined as the presence of an angiographically severe (≥70%) lesion other than the CL either proximal or distal to it in the same coronary artery after the distal flow was observed most commonly as a result of guide-wire passage or PTCA of the total occlusion.

Exclusion criteria: - Presence of LMCA lesion

* Cardiogenic shock
* Previous CABG operation
* Decision for CABG operation after primary PCI
* Severe valvular disease including aortic stenosis of mitral insufficiency
* Severe kidney disease (serum creatinine >2.5 mg/dl or patients on maintenance hemodialysis)
* Rejection of second PCI by the patient after the index event

The eligible patients were retrospectively sought from the database of the relevant hospital. The basal characteristics of the patients like age, sex, presence of coronary risk factors (smoking, hypertension, diabetes mellitus and hyperlipidemia), vital signs and location of STEMI at admission were noted. The emergent coronary angiograms of the patients were then examined and several angiographic and post-PCI features which are defined in detail in the following sections were addressed. Follow-up of these patients were succeeded either by phone call, routine polyclinic visits or from the database of hospital.

Study groups: Patients were grouped into 2 according to the PCI strategy; culprit vessel (CV) group including patients who underwent emergent PCI of all severe (≥70 stenosis in CAG) lesions in the culprit vessel and culprit lesion (CL) group including patients who underwent emergency PCI only for the CL and staged PCI in 2 weeks for the other additional lesions in the CV. Both groups underwent staged PCI for the severe lesion(s) in non-culprit vessel(s) if necessary in a different session in 28 days after the index event. Staged PCI was the preferred strategy in both groups if necessary because staged PCI has been found to be at least non-inferior to other strategies in several studies [3, 4, 10, 13].

Definition of acute STEMI: The criteria for diagnosis of STEMI were: (1) chest pain within 24 h before admission that lasted for more than 30 min and was not relieved by sublingual nitroglycerin; (2) ST-segment elevation on electrocardiogram; and (3) elevated serum creatine kinase (CK) or troponin levels.

Emergent coronary angiography and PCI procedure: All patients were routinely treated with heparin, clopidogrel, aspirin, statin and an angiotensin converting enzyme inhibitor or angiotensin II receptor blocker unless contraindicated.

Coronary angioplasty and stent implantation were performed according to standard percutaneous techniques through the femoral artery. Standard selective coronary angiography with at least 4 views of the left coronary system and 2 views of the right coronary artery was performed using the Judgkins technique.

All the patients with the diagnosis of acute STEMI underwent emergent PCI with bare metal or drug-eluting stents. Stent implantation was performed at an inflation pressure of 10 to 16 atm. When suboptimal stent deployment was observed, angiographic optimization was performed using high-pressure noncompliant balloon dilatation to achieve <20% residual stenosis by visual estimation. Angiographic no-reflow phenomenon was diagnosed if a significant coronary flow decrease (Thrombolysis In Myocardial Infarction [TIMI] grade <3 flow) without mechanical obstruction was noticed in final cineangiograms obtained at completion of the PCI procedure [14, 15].

Staged PCI: Staged PCI procedure was performed either to the culprit vessel in CL group and/or to the non-culprit lesion(s) in non-culprit vessel(s) in both groups in 14 days after the index event. In the CL group, it was performed to culprit and non-culprit vessels during same intervention. In the CV group, it was performed to non-culprit vessels if necessary.

Follow-up of patients: The investigators collected follow-up information from the database of the hospitals and/or during telephone calls with patients. Follow-up included screening for major outcomes including death (in-hospital, cardiac and non-cardiac), non-fatal myocardial infarction, and need for surgical or percutaneous revas¬cularisation.

Myocardial infarction was defined as a troponin level above the 99th percentile and symptoms of cardiac ischemia. For patients with re-infarction, the definition required ≥20% increase of cardiac markers (Troponin) with ischemic symptoms or ECG findings or angiographic evidence of coronary artery occlusion including early stent thrombosis. Early stent thrombosis was defined as acute myocardial infarction due to stent thrombosis in 30 days after implantation, usually during index hospitalization.

Statistical analysis: The analysis of the results was performed using the Predictive Analytics SoftWare (PASW) Statistics 18.0 for Windows (Statistical Package for the Social Sciences, SPSS Inc., Chicago, Illinois). Data were tested for a normal distribution using the Kolmogorov-Smirnov test. The categorical variables were shown as numbers of cases with percentages and the normally distributed continuous variables were shown as mean ± SD. Student's t-test was used for the analysis of the continuous variables that were normally distributed and the χ2 test for the categorical variables. The Kruskal-Wallis rank-sum test was used for the variables that were not normally distributed. Statistical significance was defined as p value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent primary PCI for acute STEMI and had >1 lesion in the culprit artery

Exclusion Criteria:

* Presence of LMCA lesion
* Cardiogenic shock
* Previous CABG operation
* Decision for CABG operation after primary PCI
* Severe valvular disease including aortic stenosis of mitral insufficiency
* Severe kidney disease (serum creatinine >2.5 mg/dl or patients on maintenance hemodialysis)
* Rejection of second PCI by the patient after the index event

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multi-centre retrospective study included patients from 3 high-volume primary PCI centres in Turkey. A total number of 5512 patients underwent emergent PCI for acute STEMI between January 2011 and December 2013. From this patient population, patients were looked for the presence of an additional lesion to the culprit lesion (CL). Additional lesion was defined as the presence of an angiographically severe (≥70%) lesion other than the CL either proximal or distal to it in the same coronary artery after the distal flow was observed most commonly as a result of guide-wire passage or PTCA of the total occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
MACE | 18 months